CLINICAL TRIAL: NCT00827450
Title: Effects of Coffees With Various Compositions of Antioxidants on Hepatic Steatosis Induced by a High Fructose, Hypercaloric Diet
Brief Title: Effects of Coffee on Hepatic Steatosis Induced by a High Fructose Diet
Acronym: COLIBRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Nestlé Research Center, Vers-chez-les-blanc, Switzerland (Unknown)
Responsible Party: Principal Investigator, Luc Tappy, MD, professor of physiology, University of Lausanne
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COLIBRI
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Hepatic Steatosis
Keywords: hepatic steatosis; coffee; fructose; lipids
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ctl (Placebo Comparator): control isocaloric diet; no coffee
  Interventions: Dietary Supplement: Ctl
- HF (Placebo Comparator): Hypercaloric. high fructose diet; no coffee
  Interventions: Dietary Supplement: High fructose diet; no coffee
- C1 (Experimental): Hypercaloric, high fructose diet; caffeine-free, torrefied coffee
  Interventions: Dietary Supplement: fully torrefied, caffeine-free coffee
- C2 (Experimental): Hypercaloric, high fructose diet; caffeine-free, partially torrefied coffee
  Interventions: Dietary Supplement: partially torrefied, caffeine-free coffee
- C3 (Experimental): Hypercaloric, high fructose diet; caffeinated, partially torrefied coffee
  Interventions: Dietary Supplement: Partially torrefied, caffeinated coffee

INTERVENTIONS:
Dietary Supplement: Ctl — Control, isocaloric diet; no coffee
  Arms: Ctl
Dietary Supplement: High fructose diet; no coffee — Hypercaloric, high fructose diet; no coffee
  Arms: HF
Dietary Supplement: fully torrefied, caffeine-free coffee — Hypercaloric, high fructose diet + coffee
  Arms: C1
Dietary Supplement: partially torrefied, caffeine-free coffee — Hypercaloric, high fructose diet + coffee
  Arms: C2
Dietary Supplement: Partially torrefied, caffeinated coffee — Hypercaloric, high fructose diet + coffee
  Arms: C3

SUMMARY:
This study will assess

* whether coffee consumption protects against fructose-induced hepatic steatosis in healthy humans
* whether the protective effect of coffee is dependent on it's antioxidant composition

DETAILED DESCRIPTION:
Epidemiological studies suggest that coffee consumption improves glucose homeostasis in insulin resistant subjects. An increase in intrahepatic lipids (hepatic steatosis) is highly prevalent in patients with the metabolic syndrome and may be used as a marker of altered hepatic lipid metabolism. Such an increased hepatic lipids content can be experimentally produced in healthy humans by a 6-day high fructose diet.

The purpose of this study is to evaluate whether coffee prevents hepatic lipid deposition in healthy male subjects fed a fructose-rich hypercaloric diet. Both caffeine and antioxidants (yet unspecified) may be involved.. To sort out the role of caffeine and antioxidants, we will test 3 different soluble coffee, ie fully torrefied decaffeinated coffee , partially torrefied decaffeinated coffee, and partially torrefied caffeinated coffee.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 15 kg/m2
* less than 30 min physical activity /day
* habitual coffee consumption less than three cupy /day
* consumption of caffeine-containing sodas less than 2 servings/day
* non-smoker

Exclusion Criteria:

* consumption of alcohol more than 40g/day
* presence of metallic foreign bodies
* history of eye surgery
* family history of diabetes mellitus
* history of food intolerance
* vegetarians

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
intra-hepatocellular lipid (IHCL) concentration | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement

SECONDARY OUTCOMES:
fasting plasma triglycerides | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement
fasting net lipid oxidation | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement
fasting net carbohydrate oxidation | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement
whole body ketone bodies turnover and oxidation (13C 3-hydroxybutyrate) | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement
whole body glucose turnover (6,6 2H2 glucose) | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement
whole body glycerol turnover (2H5 glycerol) | will be measured after 6 days on a hypercaloric, high fructose (4g/kg body weight/day) diet +/- treatement

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — Department of Physiology, University of Lausanne, Switzerland
Locations (1):
- Centre d'investigations cliniques "cardiomet"/ CHUV, Lausanne, Switzerland

REFERENCES:
- [Derived] Lecoultre V, Carrel G, Egli L, Binnert C, Boss A, MacMillan EL, Kreis R, Boesch C, Darimont C, Tappy L. Coffee consumption attenuates short-term fructose-induced liver insulin resistance in healthy men. Am J Clin Nutr. 2014 Feb;99(2):268-75. doi: 10.3945/ajcn.113.069526. Epub 2013 Nov 20. PMID 24257718